CLINICAL TRIAL: NCT04544839
Title: Evaluation of Patient Reported Outcome Measures and Clinical Performance of Implant Supported Overdentures With Two Different Attachment Systems: A Randomized Cross Over Clinical Study
Brief Title: Clinical Evaluation of Two Different Attachment System
Acronym: ADLCvsLOC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MCES/EC/613/2020
Record Dates: First submitted 2020-08-26; First posted 2020-09-10 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Dental Implant

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ADLC attachment in first phase (Experimental): Each patient will receive 2 implants in the canine region. Three months later, each patient will be randomized and half of the patients will receive first the ADLC (test) device (first phase). In the second phase of the crossover trial (6 months after the start of the first phase), the attachments will be replaced. Patients previously allocated to the ADLC group will receive the LOC attachments.
  Interventions: Device: ADLC attachment system with PEEK inserts
- LOC attachment in first phase (Active Comparator): Each patient will receive 2 implants in the canine region. Three months later, each patient will be randomized and half of the patients will receive first the LOC (control) device (first phase). In the second phase of the crossover trial (6 months after the start of the first phase), the attachments will be replaced. Patients previously allocated to the LOC group will receive the ADLC attachments.
  Interventions: Device: ADLC attachment system with PEEK inserts

INTERVENTIONS:
Device: ADLC attachment system with PEEK inserts — Each patient will receive 2 implants in the canine region using a guided-surgery protocol and a pre-prepared surgical stent. A healing abutment of an adequate size will be placed on the implant for transmucosal healing. The flaps will be subsequently sutured around the healing abutments. Patients' existing prostheses will be adjusted. Suture removal will be performed one week post implant placement.
  Three months later, implant level impressions will be made using the open tray technique. Each patient will be then be randomized using eCRF (electronic Case Report Form) to either ADLC group or LOC group. A final cast of the patients will be obtained and the attachments will be installed using an in-direct technique by a calibrated prosthodontists.
  Other Names: NOVALOC

SUMMARY:
Edentulous patients commonly experience a deterioration in the quality of life; both in terms of oral and general health. Studies demonstrated that conventional dentures do not adequately restore masticatory function nor quality of life. In contrast, implant-supported overdentures are considered the standard of care for edentulous patients as they offer a more stable prosthesis that ultimately results in improved oral function and patient satisfaction.

Precision attachments such as studs, magnets, telescopic crowns or a bars are commonly used for implant supported overdentures. Implant overdentures supported by stud attachments gained popularity for the rehabilitation of edentulous patients as they are self-aligning, offer dual retention and compensate for divergence between implants up to angles of 40 degrees.

However, it has been documented that the stud attachment system (Locators) requires a high frequency of maintenance, particularly with regard to the replacement of the matrix.

In order to overcome some of these limitations of existing attachment systems, a newer system was developed consisting of a matrix made of polyetheretherketone (PEEK) instead of a polymeric material. This system has an amorphous diamond like carbon-based abutment coating (ADLC) and it was claimed to be more resistant to wear.

Clinically and in vitro, no comparative studies have been performed addressing wear and retention of the traditional stud attachment and the newer ADLC attachment.

Thus, the aim of the present study is to clinically and in vitro evaluate the ADLC and study attachment system.

ELIGIBILITY:
Inclusion Criteria:

* Fully edentulous patients encountering problems (functional, aesthetics) with existing dentures in the upper and lower jaw or patients seeking for implant-supported prostheses
* Adequate bone in the anterior mandible for the placement of implants (Regular diameter implant with a minimal length of 10mm) in the canine region
* Written informed consent
* Ability to understand the procedure and to answer a questionnaire.

Exclusion Criteria:

* Impaired cognitive function and/or manual dexterity
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Unable to attend follow-up examinations
* Known or suspected non-compliance, drug or alcohol abuse
* Presence of any uncontrolled systematic disease that could compromise implant surgery and implant long-term performance
* History of radiotherapy in the head and neck region
* Heavy smoker (>10 cig. /day
* Any potential allergies or hypersensitivity to chemical ingredients of material used

  * Bruxism
  * Presence of bone metabolic disorders (e.g. osteoporosis)
  * Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2020-11-02 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Patient reported outcome measure | After a functional period of 6 months
  Mean VAS scores (visual analogue scale (0-100)) related to patient overall satisfaction for the ADLC and the LOC (Locator) attachment system provided by the patients

SECONDARY OUTCOMES:
Patient-Reported Outcome Measures (PROMs): VAS | 6 months, 1, 3, 5 years after the evaluation period of the second attachment systems
  VAS scores (visual analogue scale (0-100)) based questionnaires about retention, stability of the prosthesis, maintenance of oral hygiene, ability to speak, comfort and aesthetics will be evaluated at screening
Patient-Reported Outcome Measures (PROMs): OHIP-14 | 6 months, 1, 3, 5 years after the evaluation period of the second attachment systems
  OHIP-14 (Oral Health Impact Profile) will be evaluated at screening (Questionnaire)
Patient-Reported Outcome Measures (PROMs): Costs | 6 months, 1, 3, 5 years after the evaluation period of the second attachment systems
  Costs (INR) related to the entire treatment including additional appointments scheduled for repair and/or replacement of prostheses/matrix/matrix components
Technical outcomes: | 6 months after the first and the second evaluation period, respectively
  Questionnaire (Wear of the polymeric and PEEK inserts, Deterioration of the PEEK and polymeric inserts, Initial and final retention of the two attachment systems)
Clinical outcomes: PCR | after a functional period of 6 months for each attachment system; and1, 3 and 5 years after the evaluation period of the second attachment systems
  Plaque control record (PCR) (Questionnaire: 0/1)
Clinical outcomes: BOP | after a functional period of 6 months for each attachment system; and1, 3 and 5 years after the evaluation period of the second attachment systems
  Bleeding on probing (BOP) (Questionnaire: 0/1)
Clinical outcomes: PD | after a functional period of 6 months for each attachment system; and1, 3 and 5 years after the evaluation period of the second attachment systems
  Probing depth (PD) (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Mohit Kheur, Prof., Principal Investigator — M.A.Rangoonwala College of Dental Sciences & Research Center
Locations (1):
- M.A.Rangoonwala College of Dental Sciences & Research Center, Pune, India